CLINICAL TRIAL: NCT02740946
Title: Enhanced Function and Quality of Life Following 5 Months of Exercise Therapy for Patients With Irreparable Rotator Cuff Tears - an Intervention Study
Brief Title: Enhanced Function and Quality of Life Following 5 Months of Exercise Therapy for Patients With Rotator Cuff Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-20120040
Record Dates: First submitted 2016-04-05; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Full Thickness Rotator Cuff Tear
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise therapy (Experimental): Exercise therapy 5 months
  Interventions: Other: Exercise therapy

INTERVENTIONS:
Other: Exercise therapy — 5 months of exercise therapy with two strengthening exercises focusing on m. deltoideus anterior and m. teres minor. Furthermore, a warm up exercise was applied.

SUMMARY:
This study aims to evaluate the effect of 5 months of exercise therapy for patients with irreparable rotator cuff tears.

DETAILED DESCRIPTION:
All included patients will receive exercise therapy consisting of two exercises focusing on strengthening m. deltoideus anterior and m. teres minor.

ELIGIBILITY:
Inclusion Criteria:

* symptoms of rotator cuff rupture for at least three months with rupture of minimum musculus supraspinatus and musculus infraspinatus visualized by ultrasonography or arthroscopy
* no neurological conditions which could affect muscle strength or activity
* able to read and understand Danish
* both patients with and without a history of shoulder trauma were included

Exclusion Criteria:

* former rotator cuff surgery
* history of shoulder fracture or inflammatory conditions in the shoulder
* significant osteoarthritic changes on antero-posterior and/or lateral (outlet view) radiographs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Oxford Shoulder Score | Baseline, 3 months and 5 months
  Change is measured from baseline to 3 and 5 months

SECONDARY OUTCOMES:
EuroQuol 5 Dimensions 5 Level EQ-5D-5L | baseline and 5 months
  Change is measured from baseline to 5 months
Range of motion | Baseline and 5 months
  Range of motion measured in flexion, abduction and external rotation using a goniometer. Change is measured from baseline to 5 months
Strength | Baseline and 5 months
  Strength was measured in flexion, abduction, internal and external rotation using af dynamometer. Change is measured from baseline to 5 months
Dynamic flexion in degrees from 0 to 180 | Baseline and 5 months
  Change is measured from baseline to 5 months
Muscle activity using surface electromyography | Baseline and 5 months
  Muscle activity was measured using surface electromyography of m. trapezius superior and m. deltoideus anterior Change is measured from baseline to5 months
Pain | Baseline and 5 months
  Furthermore, patients were asked to evaluate their pain on a Visual Analogue Scale while performing flexion

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rasmussen, MD, PhD, Principal Investigator — Northern Orthopaedic Division, Aalborg University Hospital
Locations (1):
- Northern Orthopaedic Division, Aalborg University Hospital, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Christensen BH, Andersen KS, Rasmussen S, Andreasen EL, Nielsen LM, Jensen SL. Enhanced function and quality of life following 5 months of exercise therapy for patients with irreparable rotator cuff tears - an intervention study. BMC Musculoskelet Disord. 2016 Jun 8;17:252. doi: 10.1186/s12891-016-1116-6. PMID 27278468